CLINICAL TRIAL: NCT02315105
Title: Resolution of Comorbidities & Safety and Efficacy of Greater Curvature Plication in Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singh, Kuldeep, M.D., P.A. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT0151290
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Morbid Obese patients (Experimental): This purpose of this study is to find out more about the safety and effectiveness of the Laparoscopic Greater Curvature Plication (LGCP) for Morbid Obese Patients with related problems such as diabetes, hypertension, high cholesterol, mild obstructive sleep apnea and joint problems.
  Interventions: Procedure: Laparoscopic Greater Curvature Plication

INTERVENTIONS:
Procedure: Laparoscopic Greater Curvature Plication — LGCP is a procedure in which the stomach is folded inwards to that its capacity to hold amount of food is decreased dramatically. This is done under general anesthesia. The operation takes about 1 hour and is done laparoscopically. The attachments of the stomach to the spleen are feed up and the outside is folded inside and stitched up to keep it from folding in. To ensure that the surgeon has not obstructed the passage in or out of the stomach, a tube ( Bougie) is placed in the stomach at the time of the creation of the fold and checked again at the end of the procedure with a camera in the stomach which is placed through the mouth (EGD- upper endoscopy) to ensure the desired outcome is achieved.

SUMMARY:
The purpose of this study is to find out more about the safety and effectiveness of the Laparoscopic Greater Curvature Plication (LGCP) procedure in patients with obesity and related problems such as diabetes, hypertension, high cholesterol, mild obstructive sleep apnea, and joint problems. LGCP is a less invasive weight loss surgery procedure than some of the other weight loss surgeries and it is possible that there are fewer risks with this procedure than with the other weight loss surgeries. LGCP is considered an experimental procedure and this study is being done to look at the long-term outcomes.

DETAILED DESCRIPTION:
LGCP is a procedure in which the stomach is folded inwards to that its capacity to hold amounts of food is decreased. This is done under general anesthesia. The operation takes about an hour and is done laparoscopically. Laparoscopic approach entails placing 4-5 small incisions in the abdomen around the umbilicus and filling the abdomen with CO2 through the small tubes called Trocars. this helps life the abdominal wall and create space so that the surgeon can carry out his/her work using long instruments with thickness similar to a regular lead pencil.

The attachments of the stomach to the spleen are freed up and the outside is folded inside and stitched up to keep it from folding in. To ensure that the surgeon has not obstructed the passage in or out of the stomach, a tube is placed in the stomach at the time of the creation of the fold and checked again at the end of the procedure with a camera in the stomach which is placed through the mouth to ensure the desired outcome is achieved. At the conclusion of the procedure, the skin is closed with absorbable sutures and adhesive tapes are applied to the skin. The patient recovers in the recovery room for about an hour and a half prior to coming to their room in the hospital.

The post operative visit will be up to 7 days after the procedure. During this visit, medical information will be obtained including information about medications.

There will be follows 3-10 after the surgery. These visits may include:

* obtaining medical information about the patient, including the medical conditions and medications
* Checking the patient's weight
* Blood tests
* Endoscopic evaluation of the stomach if necessary.

The timing of the visits is as follows:

Visit 3: 1 month after surgery Visit 4: 3 months after surgery Visit 5: 6 months after surgery Visit 6: 12 months after surgery Visit 7: 18 months after surgery Visit 8: 24 months after surgery Visit 9: 30 months after surgery Visit 10: 36 months after surgery

The study is three (3) years (36 months) including following up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing to give consent and comply with evaluation and treatment schedule
2. 18 to 65 years of age
3. Have a BMI > 30 with one or more significant co-morbid medical conditions which are generally expected to be improved, reversed, or resolved by weight loss. these conditions include but are not limited to:

   * Hyperlipidemia
   * Type 2 diabetes
   * Mild Obstructive Sleep Apnea
   * Hypertension
   * Osteoarthritis of the hip or knee
4. Agree to refrain from any type of weight-loss drug ( prescription or OTC) or elective procedure that would affect body weight for the duration of the trial
5. HbA1C < 11 %
6. For subjects who have Type 2 Diabetes, the anti-diabetic medication regimen is no more complex than oral metformin plus one oral sulfonylurea plus once daily insulin injection.
7. Ability to self-pay for the procedure and follow up.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Percent excess weight loss | 1 year

SECONDARY OUTCOMES:
Resolution of Comorbidities | 1 year
  After one year, evaluate each patient to see if the patient has had resolution of any types of comorbidities they manifested pre op; diabetes, hypertension, high cholesterol, mild obstructive sleep apnea, and joint problems

CONTACTS AND LOCATIONS:
Overall Officials: Kuldeep Singh, MD, Principal Investigator — Saint Agnes Hospital
Locations (1):
- Saint Agnes Hospital, Baltimore, Maryland, United States